CLINICAL TRIAL: NCT02837640
Title: The Effect of L-Dopa on the Progression of Retinitis Pigmentosa
Brief Title: Studying a Potential Protective Effect of L-Dopa on Retinitis Pigmentosa
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beirut Eye Specialist Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RP DOPA
Record Dates: First submitted 2016-06-22; First posted 2016-07-19 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2016-07

CONDITIONS: Retinitis Pigmentosa
Keywords: Retinitis Pigmentosa; Levodopa
MeSH Terms: conditions — Retinitis Pigmentosa | interventions — carbidopa, levodopa drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): This is a single armed study. All patients included will receive treatment. Control will happen with data from the same patients before they received treatment.
  patients will receive sinemet 200/50 1/2 tablet (levodopa-carbidopa 100/25) b.i.d for two days and then will be increased to t.i.d. for 6 months.
  Interventions: Drug: levodopa-carbidopa

INTERVENTIONS:
Drug: levodopa-carbidopa — sinemet 200/50 1/2 tablet b.i.d. for 2 days and then t.i.d for 6 months
  Other Names: Sinemet 200/50

SUMMARY:
The purpose of this study is to evaluate the effect of L-Dopa on the progression of retinitis pigmentosa.

DETAILED DESCRIPTION:
Retinitis pigmentosa is a group of progressive hereditary diseases that diffusely affects the functioning of photoreceptors and the pigment epithelium. It may be speculated that a protective effect on the pigment epithelium, as it is supposed for L-Dopa, can slow the progression of the disease or even lead to an, at least transient, improvement of visual functions. To evaluate the effect of L-Dopa on retinitis pigmentosa progression, visual acuity, electroretinogram and visual field will be preformed regularly.

ELIGIBILITY:
Inclusion Criteria:

* All confirmed cases of retinitis pigmentosa
* VA of 20/400 or better

Exclusion Criteria:

* Advanced stages of retinitis pigmentosa with poor best corrected visual acuity (less than 20/400)
* co-existing eye morbidities interfering with retinitis pigmentosa (glaucoma, retinal detachment...)
* Flat electroretinogram
* Intolerance or counterindication to drug
* Unability for long-term follow-up

Ages: 10 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Change in Electroretinogram | Baseline, 1 year, 2 years, 5 years
  the electric response to light stimuli of the retina, in millivolt, will be measured. The electroretinogram shows a-waves (elicit information about the function of the photoreceptors) and b-waves (elicit information about other neurosensory structure of the retina)

SECONDARY OUTCOMES:
Change in Visual Acuity | Baseline, 6 months, 1 year, 2 years, 5 years
  Visual acuity will be measured using Snellen chart
Change in Visual Field | Baseline, 1 year, 2 years, 5 years
  Using 24-2 Humphrey Visual Field Analyzer, the progress in visual field defect will be measured, comparing mean deviation (dB) and pattern standard deviation (dB)

CONTACTS AND LOCATIONS:
Overall Officials: Elias F. Jarade, MD, Principal Investigator — Beirut Eye Specialist Hospital
Locations (1):
- Beirut Eye Specialist Hospital, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: No
Individual participant date will not be shared at the moment being, since it is not of value unless it is thoroughly analysed.

REFERENCES:
- [Background] Brilliant MH, Vaziri K, Connor TB Jr, Schwartz SG, Carroll JJ, McCarty CA, Schrodi SJ, Hebbring SJ, Kishor KS, Flynn HW Jr, Moshfeghi AA, Moshfeghi DM, Fini ME, McKay BS. Mining Retrospective Data for Virtual Prospective Drug Repurposing: L-DOPA and Age-related Macular Degeneration. Am J Med. 2016 Mar;129(3):292-8. doi: 10.1016/j.amjmed.2015.10.015. Epub 2015 Oct 30. PMID 26524704